CLINICAL TRIAL: NCT03995095
Title: Intervention in Spirituality at the End of Life. The Kibo Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Sociedad Española de Cuidados Paliativos SECPAL (Unknown)
Responsible Party: Principal Investigator, M. Antonia Pérez-Marín, Profesora Titular, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H1447334931417
Record Dates: First submitted 2019-06-05; First posted 2019-06-21 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Palliative Care
Keywords: Spirituality; Intervention Study

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Group of participants that received usual psychological attention.
- Experimental group (Experimental): Group of participants that received usual psychological attention plus attention of spiritual needs following the Kibo protocol (intervention).
  Interventions: Other: Therapeutic interview: kibo protocol

INTERVENTIONS:
Other: Therapeutic interview: kibo protocol — The kibo protocol is a therapeutic interview designed to address the spiritual needs of patients at the end of life.
  Arms: Experimental group

SUMMARY:
This work aims to study the benefits that the therapeutic interview Kibo in palliative care patients can have for spirituality.

A parallel randomized controlled trial of two groups was performed. Information was collected on 60 palliative care patients during the moments before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. To be 18 or more years of age.
2. Being in advanced or terminal disease phase (following World Health Organization criteria).
3. To have preserved cognitive capacity.
4. To have signed the informed consent.

Exclusion Criteria:

a) Estimated time of survival: Patients with a life expectancy of two weeks or less will not be intervened.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in the dimension of spirituality (PRE and POST measures) | Baseline up to 4 weeks
  This variable was assessed with the Spirituality questionnaire from the Spanish Society of Palliative Care (SECPAL). This questionnaire contains 8 items, and it provides scores from 0 to 32, where higher values represent a better outcome.
  In order to observe the change in the dimension of spirituality, it was measured at in two time points:
  First measurement: PRE. Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: POST. Up to 4 weeks after the first measurement, the second measurement of the same variable was carried out.
  Between first and second measurement, the control group received the usual psychological attention, whereas the intervention group received usual psychological attention plus attention of spiritual needs following the Kibo protocol (intervention).

SECONDARY OUTCOMES:
Change in resilience (PRE and POST measures) | Baseline up to 4 weeks
  This variable was assessed with the Brief Resilient Coping Scale (BRCS). This scale contains 4 items, and it provides scores from 4 to 20, where higher values represent a better outcome.
  In order to observe the change in the dimension of resilience, it was measured at in two time points:
  First measurement: PRE. Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: POST. Up to 4 weeks after the first measurement, the second measurement of the same variable was carried out.
  Between first and second measurement, the control group received the usual psychological attention, whereas the intervention group received usual psychological attention plus attention of spiritual needs following the Kibo protocol (intervention).
Change in demoralization (PRE and POST measures) | Baseline up to 4 weeks
  This variable was assessed with the Short Demoralization Scale (SDS). This scale contains 5 items, and it provides scores from 0 to 20, where lower values represent a better outcome.
  In order to observe the change in the dimension of demoralization, it was measured at in two time points:
  First measurement: PRE. Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: POST. Up to 4 weeks after the first measurement, the second measurement of the same variable was carried out.
  Between first and second measurement, the control group received the usual psychological attention, whereas the intervention group received usual psychological attention plus attention of spiritual needs following the Kibo protocol (intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Barreto Martin, PhD, Principal Investigator — Universitat de València
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soto-Rubio A, Perez-Marin M, Rudilla D, Galiana L, Oliver A, Fombuena M, Barreto P. Responding to the Spiritual Needs of Palliative Care Patients: A Randomized Controlled Trial to Test the Effectiveness of the Kibo Therapeutic Interview. Front Psychol. 2020 Aug 21;11:1979. doi: 10.3389/fpsyg.2020.01979. eCollection 2020. PMID 32973614